CLINICAL TRIAL: NCT00824720
Title: Safety and Efficacy of a Glaucoma Drug Delivery System
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Vistakon Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR-1630
Record Dates: First submitted 2009-01-09; First posted 2009-01-19 (Estimated); Results first posted 2010-05-14 (Estimated); Last update posted 2015-03-06 (Estimated); Status verified 2015-02

CONDITIONS: Glaucoma, Open-Angle; Ocular Hypertension
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- High Dose Device (Experimental): device worn continuously for 14 days
  Interventions: Drug: High Dose Device
- Low Dose Device (Experimental): device worn continuously for 14 days
  Interventions: Drug: Low Dose Device
- Placebo Device (Placebo Comparator): device worn continuously for 14 days
  Interventions: Device: Placebo Device

INTERVENTIONS:
Drug: High Dose Device — inserted for 14 days
  Arms: High Dose Device
Drug: Low Dose Device — inserted for 14 days
  Arms: Low Dose Device
Device: Placebo Device — inserted for 14 days
  Arms: Placebo Device

SUMMARY:
The purpose of this study is to evaluate the ocular safety and efficacy of a glaucoma drug delivery system in open-angle glaucoma or ocular hypertension.

ELIGIBILITY:
Inclusion Criteria:

* Man or woman 21 years of age or greater
* must have open angle glaucoma or ocular hypertension.
* Corrected visual acuity in each eye of 20/200 or better.

Exclusion Criteria:

* Previous glaucoma intraocular surgery or refractive surgery.
* Planned contact lens use during the study.
* Clinically significant ocular or systemic disease that might interfere with the study.
* Use of chronic corticosteroids by any route.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2008-12; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Artesia, California
  - Louisville, Kentucky
  - Baltimore, Maryland
  - Mt. Pleasant, South Carolina

RESULTS

PARTICIPANT FLOW:
Groups:
- High Dose Bimatoprost Punctal Plug: punctal plug with bimatoprost, high dose
- Low Dose Bimatoprost Punctal Plug: punctal plug with bimatoprost, low dose
- Placebo: punctal plug without bimatoprost
Period: Overall Study
Arm/Group | High Dose Bimatoprost Punctal Plug | Low Dose Bimatoprost Punctal Plug | Placebo
Started | 19 (3 subjects in the high dose group did not receive device - unable to insert.) | 16 (1 subject in the low dose group did not receive device - unable to insert.) | 20
Completed | 16 | 15 | 19
Not Completed | 3 | 1 | 1
Not completed — failed plug insertion | 3 | 1 | 0
Not completed — Protocol Violation | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | High Dose Bimatoprost Punctal Plug | Low Dose Bimatoprost Punctal Plug | Placebo | Total
Number analyzed (Participants) | 16 | 15 | 20 | 51
Age, Continuous [Mean (Standard Deviation); unit: years] — This baseline measure includes all subjects with a plug insertion.
  years | 66.7 (13.4) | 64.6 (12.9) | 64.5 (10.6) | 65.2 (12.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 9 | 13 | 31
  Male | 7 | 6 | 7 | 20

OUTCOME MEASURES:

1. Secondary Outcome: Intraocular Pressure (IOP)
Time Frame: from baseline to 14 days
Population: The analysis population includes all subjects with a plug insertion that completed the study per protocol.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | High Dose Bimatoprost Punctal Plug | Low Dose Bimatoprost Punctal Plug | Placebo
Number analyzed (Participants) | 14 | 15 | 19
mmHg | -1.9 (2.3) | -2.2 (3.5) | -1.3 (3.6)
Statistical Analysis 1: Comparison: High Dose Bimatoprost Punctal Plug vs Placebo; The alternative hypothesis was that the high dose was different from the placebo; Test type: Superiority or Other; p = 0.9737, ANCOVA; least square mean difference = -0.22, Standard Deviation 2.3 — Mean difference was calculated as high dose minus placebo
Statistical Analysis 2: Comparison: Low Dose Bimatoprost Punctal Plug vs Placebo; The alternative hypothesis is that the low dose was different from placebo; Test type: Superiority or Other; p = 0.4711, ANCOVA; least square mean difference = -1.11, Standard Deviation 3.5 — The mean difference was calculated as low dose minus placebo

2. Primary Outcome: Visual Acuity - Right Eye
Description: This outcome measures visual acuity in logMARs. logMAR is the logarithm of the minimum angle of resolution (logMAR). The ideal is 0.0 and represents 20/20 Snellen acuity. logMar values > 0.00 indicate vision poorer than the ideal and values <0.00 indicate vision greater than the ideal.
Time Frame: at 14 days
Measure: Mean (Standard Deviation); unit: logMAR units
Arm/Group | High Dose Bimatoprost Punctal Plug | Low Dose Bimatoprost Punctal Plug | Placebo
Number analyzed (Participants) | 14 | 15 | 19
logMAR units | 0.015 (0.046) | -0.044 (0.092) | -0.012 (0.044)

3. Primary Outcome: Visual Acuity - Left Eye
Description: This outcome measures visual acuity in logMARs. logMAR is the logarithm of the minimum angle of resolution (logMAR. The ideal is 0.0 and represents 20/20 Snellen acuity. logMar values > 0.00 indicate vision poorer than the ideal and values <0.00 indicate vision greater than the ideal.
Time Frame: at 14 days
Measure: Mean (Standard Deviation); unit: logMARs
Arm/Group | High Dose Bimatoprost Punctal Plug | Low Dose Bimatoprost Punctal Plug | Placebo
Number analyzed (Participants) | 14 | 15 | 19
logMARs | -0.011 (0.081) | -0.008 (0.101) | -0.019 (0.044)

ADVERSE EVENTS:
Arm/Group | High Dose Bimatoprost Punctal Plug | Low Dose Bimatoprost Punctal Plug | Placebo
Serious Adverse Events (participants affected / at risk) | 1/16 | 0/15 | 0/20
Other Adverse Events (participants affected / at risk) | 13/16 | 11/15 | 11/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | High Dose Bimatoprost Punctal Plug (N=16) | Low Dose Bimatoprost Punctal Plug (N=15) | Placebo (N=20)
cerebrovascular accident (Nervous system disorders) | 1 | 0 | 0 — unrelated to study treatment
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | High Dose Bimatoprost Punctal Plug (N=16) | Low Dose Bimatoprost Punctal Plug (N=15) | Placebo (N=20)
Foreign body sensation (Eye disorders) | 8 | 5 | 3
Eye pain (Eye disorders) | 6 | 2 | 1
abnormal sensation in eyes (Eye disorders) | 5 | 3 | 4
Conjunctival hyperaemia (Eye disorders) | 3 | 5 | 2
corneal erosion (Eye disorders) | 5 | 2 | 0
dry eye (Eye disorders) | 3 | 2 | 0
erythema of eyelid (Eye disorders) | 1 | 0 | 0
eye irritation (Eye disorders) | 1 | 0 | 0
eye puritus (Eye disorders) | 0 | 0 | 1
eyelid margin crusting (Eye disorders) | 4 | 1 | 2
eyelid pain (Eye disorders) | 5 | 2 | 1
eyelids puritus (Eye disorders) | 0 | 0 | 1
inflammation of lacrimal passage (Eye disorders) | 5 | 4 | 2
lacrimation increased (Eye disorders) | 2 | 5 | 4
ocular hyperaemia (Eye disorders) | 3 | 2 | 0
visual acuity reduced (Eye disorders) | 0 | 0 | 1
upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0
contusion (Injury, poisoning and procedural complications) | 0 | 1 | 0
procedural complication (Injury, poisoning and procedural complications) | 1 | 0 | 2
musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
sinus headache (Nervous system disorders) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Prior to submission for publication or presentation, the PI will provide the Sponsor 60 days for review of the manuscript. The Sponsor may request that the PI withhold the publication for an additional 60 days.